CLINICAL TRIAL: NCT01512394
Title: Effects of Preoperative Bowel Preparation Prior to Elective Bowel Resection or Ostomy Closure in the Pediatric Patient Population
Brief Title: Pre-op Bowel Prep Before Abdominal Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never started.
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: University of North Carolina (Other)
Responsible Party: Principal Investigator, Shawn St. Peter, Associate Professor, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11 09-139
Record Dates: First submitted 2011-12-13; First posted 2012-01-19 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Pre-operative Bowel Prep
Keywords: bowel preparation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard bowel prep (Active Comparator): Standard bowel prep
  Interventions: Procedure: standard bowel prep
- No bowel prep (Experimental): No bowel prep
  Interventions: Procedure: no bowel prep

INTERVENTIONS:
Procedure: standard bowel prep — standard bowel prep
  Arms: Standard bowel prep
Procedure: no bowel prep — no bowel prep
  Arms: No bowel prep

SUMMARY:
Current management of elective bowel surgery typically involves performing a preoperative bowel preparation ("bowel prep") in many instances; however, this practice is not standardized at most institutions. Over the years, bowel preps have been used in an attempt to decrease the risk of complications associated with gastrointestinal surgery. However, there is limited adequate data to support this clinical management in the pediatric patient population. The investigator plans to perform a prospective, randomized study of our pediatric surgical patients who will undergo an elective bowel resection or ostomy closure to assess if a bowel prep prior to surgical intervention affects their postoperative course. The aim of this study is to evaluate for differences that may alter and improve future management.

DETAILED DESCRIPTION:
At CMH, our current approach to preoperative management for elective intestinal surgery is not standardized amongst our Pediatric Surgical attendings. There are seven different attendings, each of whom individually dictates if a patient is to undergo a preoperative bowel prep, and if so, which bowel prep will be used. This is no different than the majority of practices across the US, including adult and pediatric patient populations. The aim of this study, therefore, is to standardize our current management and assess if the presence or absence of a preoperative bowel prep has an effect on post-operative outcomes. The goal is to evaluate the effect of the bowel preparation not the surgical procedure itself.

ELIGIBILITY:
Inclusion Criteria:

* All children, ages 3 months to 17 years, who will undergo an elective bowel resection or ostomy closure at CMH

Exclusion Criteria:

* Patients whose operation was performed emergently, and hence a bowel prep was not possible preoperatively;
* If they necessitate a diverting proximal ostomy;
* If they have any known intra-abdominal infection preoperatively;
* If an intra-operative colonoscopy is necessary, and hence the patient must have a preoperative bowel prep.
* No patients with an underlying malignancy or immunodeficiency or with renal, metabolic or cardiac conditions will be included.
* No patients with known allergies to any medication used in the bowel preparation will be included.

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
complications following surgery | 6 weeks
  compications such as infection, leaks, obstruction etc

SECONDARY OUTCOMES:
Length of hospital stay | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States